CLINICAL TRIAL: NCT04702672
Title: High-amylose Barley (HIAMBA) in the Regulation and Prevention of Type 2 Diabetes: a Randomized, Cross-over, Acute Dietary Intervention Study.
Brief Title: High-amylose Barley (HIAMBA) in the Regulation and Prevention of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HIAMBA-2
Record Dates: First submitted 2020-12-09; First posted 2021-01-11 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes
Keywords: Glycemic index; Postprandial; Barley; High-amylose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, cross-over, acute, dietary intervention study
Who Masked: Participant
Masking Description: Letter labeling of test products
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetes (Experimental): Adults with T2D. Hemoglobin A1C between 42-78 mmol/l. No use of insulin or once-weekly glucagon-like peptide-1 (GLP-1) or acarbose. No severe cardiovascular, kidney, liver, psychiatric or endocrine disease. No abuse of alcohol- or narcotics. No pregnancy or lactation.
  Interventions: Dietary Supplement: 100% wheat (control); Dietary Supplement: 100% Lean-baking barley®; Dietary Supplement: 100% regular barley
- Non-diabetics (Experimental): Adults without T2D. No severe cardiovascular, kidney, liver, psychiatric or endocrine disease. No abuse of alcohol- or narcotics. No pregnancy or lactation.
  Interventions: Dietary Supplement: 100% wheat (control); Dietary Supplement: 100% Lean-baking barley®; Dietary Supplement: 100% regular barley

INTERVENTIONS:
Dietary Supplement: 100% wheat (control) — Intake of 250 ml of tap water and 100 g of bread baked with 100% wheat flour (regular commercial available wheat flour). Consumed over maximum 10 minutes at time 0 min after overnight fasting. At one of four visits.
Dietary Supplement: 100% Lean-baking barley® — Intake of 250 ml of tap water and 100 g of bread baked with 100% Lean-baking barley® flour. Consumed over maximum 10 minutes at time 0 min after overnight fasting. At one of four visits.
  HIAMBA® are naturally bred in corporation with PlantCarb ApS and researchers at Aarhus and Copenhagen Universities. The wheat flour is standard commercial available flou
Dietary Supplement: 100% regular barley — Intake of 250 ml of tap water and 100 g of bread baked with 100% regular barley flour and 25% wheat flour. Consumed over maximum 10 minutes at time 0 min after overnight fasting. At one of four visits.
  HIAMBA® are naturally bred in corporation with PlantCarb ApS and researchers at Aarhus and Copenhagen Universities. The wheat flour is standard commercial available flour.

SUMMARY:
In a series of double-blinded randomized cross-over acute studies, the investigators want to study the effects of naturally produced high-amylose barley (Lean-baking barley®) on the postprandial glucose-metabolism in subjects with and without type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The prevalence of T2D is increasing worldwide, primarily due to obesity, lack of physical activity and unhealthy diet. Therefore, it is of great important to evolve dietary products that counteracts this development.

Barley has shown some beneficial effects on postprandial blood glucose compared with wheat. A lowering of the postprandial glucose level reduces the risk of developing T2D and helps in the regulation of a pre-existing diabetes. However, barley is traditionally not used in bread-making in Denmark.

The elevation of postprandial glucose also depends on how fast the dietary products are degraded in the gastrointestinal tract.

The starch in barley consist of both fastly degraded amylopectin and slowly degraded amylose. Slow degradation is expected to lower postprandial glucose. By natural breeding techniques it has been possible for the investigators collaborative partners at the Universities of Aarhus and Copenhagen and PlantCarb ApS to make an natural organic high-amylose barley (Lean-baking barley®).

In a series of acute studies the investigators want to study the effects on the glycemic response to bread made with different flours (wheat, regular barley, Lean-baking barley® in subjects with T2D.

The investigators expect that Lean-baking barley® positively affect the postprandial glucose-metabolism more than wheat and regular barley and hereby acutely improves the glycemic regulation for both subjects with and without T2D.

ELIGIBILITY:
Inclusion Criteria for T2D group:

* T2D defined by standard Danish guidelines.
* HbA1c between 42-78 mmol/l.
* Treatment with drugs for hypertension and high cholesterol is allowed if the treatment dose is stable and does not demand changes during the study period.
* Participants are encouraged to maintain their present psychical activity level and their smoking and alcohol habits.

Exclusion Criteria:

* Type 1 diabetes
* Insulin demanding T2D
* Use of weekly administrated GLP-1 antagonist (e.g. ozempic, trulicity or byetta)
* Use of acarbose
* Significant cardiovascular, kidney, liver or endocrine comorbidity
* Significant psychiatric history
* Treatment with steroids
* Alcohol or drug abuse
* Pregnancy or breastfeeding
* Legally incompetent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response | Time Frame: Change from -10 minutes to 240 minutes after bread intake (measured at time -10,0,10,20,30,45,60,90,120,150,180,210,240 minutes)
  Postprandial glycemic response Area under the curve for glucose (mmol/L)

SECONDARY OUTCOMES:
Postprandial insulin response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,10,20,30,45,60,90,120,150,180,210,240 minutes)
  Area under the curve for insulin (pmol/L)
Postprandial glucagon response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,10,20,30,45,60,90,120,150,180,210,240 minutes)
  Area under the curve for glucagon (pg/mL)
Postprandial triglyceride response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,30,60,120,180,240 minutes)
  Area under the curve for triglyceride (mmol/L)
Postprandial free fatty acid response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,30,60,120,180,240 minutes)
  Area under the curve for free fatty acids (mmol/L)
Postprandial GLP-1 (glucagon-like peptide-1) response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,30,60,120,180,240 minutes)
  Area under the curve for GLP-1 (pmol/L)
Postprandial GIP (Glucose-dependent insulinotropic polypeptide) response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,30,60,120,180,240 minutes)
  Area under the curve for GIP (pmol/L)
Visual analogue scale (VAS) | Measured at time 0,30,60,90,120,150,180,210,240 minutes
  VAS-score of a number of standardized questions regarding, hunger, satiety, the test meal experience etc. Each answer is ranged on a 100 mm line expressing the most positive and negative rating possible at each end.

CONTACTS AND LOCATIONS:
Overall Officials: Mette B Larsen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Bohl M, Gregersen S, Li Z, Blennow A, Hebelstrup KH, Hermansen K. High-amylose barley bread improves postprandial glycemia compared to regular barley and wheat bread in subjects with or without type 2 diabetes. Eur J Clin Nutr. 2025 Oct;79(10):1000-1006. doi: 10.1038/s41430-025-01646-6. Epub 2025 Jul 21. PMID 40691269